# **Evaluating the Effect of Facilitated Enrollment and Enhanced Outreach Strategies on Marketplace Health Insurance Take-up**

Emory Wolf, MPP, Covered California 1601 Exposition Blvd Sacramento CA 95815 Emory.wolf@covered.ca.gov

Marina Lovchikova, PhD, Covered California, 1601 Exposition Blvd Sacramento CA 95815 Marina.lovchikova@covered.ca.gov

Isaac Menashe, MPP, Covered California 1601 Exposition Blvd Sacramento CA 95815 <a href="mailto:lsaac.menashe@covered.ca.gov">lsaac.menashe@covered.ca.gov</a>

Katie Ravel, MPH, Covered California 1601 Exposition Blvd Sacramento CA 95815 Katie.ravel@covered.ca.gov

Valerie York, Covered California 1601 Exposition Blvd Sacramento CA 95815 Valerie.york@covered.ca.gov

# **Funding**

None

## **Conflict of Interest**

None

Date of the document creation: May 2, 2024

# **Design Document and Analysis Plan**

# **Project Objective**

For individuals who do not have coverage through their employers or state Medicaid programs, health insurance take-up remains incomplete, despite significantly reduced premiums, and even free coverage for many of these uninsured. Facilitated enrollment offers a potential solution to some administrative burdens and choice frictions that produce this incomplete take-up of marketplace coverage. Because Covered California, California's ACA individual marketplace, and Medi-Cal, California's Medicaid program, share an eligibility system, Covered California has the ability to identify individuals who are eligible for marketplace coverage upon losing Medicaid eligibility.

This evaluation will compare the effectiveness of facilitated enrollment strategies on marketplace take-up among individuals losing Medi-Cal coverage, by comparing outcomes for personalized plan pre-selection and personalized quotes of net premiums, to other more general outreach tactics (such as reminder nudges).

# **Target population**

The study population includes single-member households who are discontinued from Medi-Cal and found eligible for Covered California. The study leverages application differences between the Medi-Cal and Covered California programs, the latter of which requires that individuals attest to plan to file taxes in order to receive premium subsidies, in the form of advanced premium tax credits (APTCs). Individuals who did not answer this question on their Medi-Cal application are found ineligible for marketplace premium subsidies when discontinued from Medi-Cal. Thus, many individuals are missing out on financial assistance that they are likely eligible for because of these discrepancies in program requirements.

The study population will focus on this subset of consumers, rerunning their program eligibility to check for subsidy eligibility after suggesting changes to the tax filing questions within the application. The exact inclusion criteria are:

- Individual in a single-member household
- Discontinued from Medi-Cal
- Eligible for Covered California program
- Ineligible for APTCs
- Did not attest to planning to file taxes within their Covered California application
- Do not meet any of the exclusion criteria:
  - o Consumer case is no longer active within the application system
  - o Consumer is already actively enrolled in a marketplace plan
  - Consumer has already restored Medi-Cal eligibility
  - o A consumer's Special Enrollment Period has ended
  - o Consumer is no longer listed as a single-member household
  - o Consumer was procedurally denied from Medi-Cal coverage due to no response
  - Consumers has a MAGI Medi-Cal income less than 138% of the Federal Poverty Level (FPL)

## Interventions and Randomization

The project's research design is a randomized intervention among single-member households who have recently lost Medi-Cal coverage, are found eligible for marketplace coverage, but are

ineligible for subsidies due to incomplete application information regarding planning to file taxes. After meeting the inclusion criteria above, individuals are randomly assigned to one of three treatment arms:

- 1. A control group that receives a standard eligibility notice informing them of their eligibility for marketplace coverage.
- 2. A treatment group that receives a standard eligibility notice informing them of their eligibility for marketplace coverage and an informational flyer describing what Covered California is, the availability of financial assistance, and information on benefit design and private insurance terminology, such as deductibles and copays.
- 3. A treatment group that receives a modified eligibility notice that includes information on the pre-selected lowest-cost silver health insurance plan with a personalized quote for their net premium amount, as well as the informational flyer.

The evaluation will run for two years and include approximately 30,000 individuals who have been discontinued from Medi-Cal coverage. An estimated 6,000 individuals will be assigned to the control and estimated 12,000 individuals will be assigned to one of the two treatment arms.

#### Power:

To arrive at an estimate for the minimum detectable effect (MDE) for our primary outcome, we assume a baseline health insurance take up of 6 percent. The baseline rate was determined with the historical data on the plan effectuation of single-member households disenrolled from Medi-Cal in 2018-2019 years. The intervention has 80% power to detect a 1.1 percentage point increase in effectuation<sup>1</sup>.

# **Likely Effect Size:**

Based on prior personalized outreach campaigns carried out by Covered California, we would expect to observe an ITT effect between 0 and 4 percentage points with lower bound point likely detected for the enhanced outreach group and upper bound detected for the treatment group with personalized quote information.

## **Data and Data Structure**

### **Outcomes:**

We use Covered California administrative data to examine health insurance take-up behavior and health care utilization among households included in the study and found eligible for premium subsidies at the time of the intervention.

The primary outcome of interest will be a binary indicator for whether a consumer has at least one month of effectuated coverage a Covered California plan within the 90 days of their Special Enrollment Period (SEP) following loss of Medi-Cal coverage.

Our secondary outcomes will be measured 1-2 years after the intervention when data becomes available will include:

- 1. Tenure with Covered California (measured in months);
- 2. A binary indicator for whether someone self-reported being uninsured while filing their taxes;

<sup>&</sup>lt;sup>1</sup> Authors' calculations based on a two-sample proportion Pearson's chi-squared test using Stata 18 SE software

- 3. A binary indicator for consumer engagement (including calls to service center, logins to user account, agent delegation after eligibility determination);
- 4. A binary indicator for whether someone had an office visit during 1-2 years since the intervention;
- 5. A binary indicator for whether someone had a prescription drug fill during 1-2 years since the intervention;
- 6. A binary indicator for whether someone had an emergency room visit during 1-2 years since the intervention:
- 7. A binary indicator for whether someone had a hospital admission 1-2 years before and during 1-2 years since the intervention.
- 8. Total out-of-pocket spending for the 1-2 years since the intervention

#### Data:

We will use Covered California administrative data to obtain enrollment outcomes and baseline demographics for our sample and Covered California's health care claims database to obtain health care utilization and financial outcomes for individuals who enroll in coverage. Administrative data from pilot months (March-May 2024) of program implementation have been reviewed to provide insight on sample size estimation. Data from these pilot months will be included in the analysis.

We will use data from the Department of Health Care Access and Information for hospital admissions data for all individuals in the intervention. We will use data from the California Franchise Tax Board to measure which individuals reported not having Minimum Essential Coverage (MEC) while filing their state taxes.

## **Quality Control Checks:**

After carrying out the randomization, we will check for balance across several observable covariates (e.g., gender, presence of email address on the application, age, race/ethnicity, language, and income as a percent of the federal poverty level), which could indicate that there would be no significant dissimilarities across treatment arms.

We will segment and separately review data collected for cases with eligibility determinations for program start dates October through December, as many of these consumers will have a different enrollment experience than the main analytic sample.

## Statistical Models

**Intention-to-treat estimation:** To estimate treatment effects, our primary analysis will be an intent-to-treat (ITT) specification, examining the effect of treatment assignment. We will estimate the effect of the treatment using ordinary least squares (OLS) regression. Covariates identified during quality control checks will be included in the model. We will regress the outcome of interest (e.g., take-up) for household *i* on the treatment indicator:

outcome; =  $\propto$ +  $\beta_1$  1(Treatment 1=1); +  $\beta_2$  1(Treatment 2= 1); +  $\epsilon_i$ 

The coefficients  $\beta_1$  and  $\beta_2$  will be the intent-to-treat estimate of the causal effect of the outreach.

**Complier average causal effect estimation:** We will examine the effects of health insurance (among households induced to enroll in a Covered California as a result of random assignment) on our four utilization outcomes. We anticipate a significant share of noncompliers among those

households assigned to receive outreach (intervention) as they may have opted out of assigned plan or not enroll into another Covered California plan. Thus, to augment our analysis of insurance take-up, we will also estimate treatment effects based on treatment receipt (enrollment into Covered California Plan), using two-stage least squares regression (2SLS).

# **Pre-Specified Subgroup Analyses**

Same subgroup analyses will be performed for our complier average causal effect analysis.

## Inference Criteria, Including Any Adjustments for Multiple Comparisons:

We will not perform any corrections for multiple hypothesis testing, and we will use two-tailed tests with p-values <= 0.05 to denote statistically significant effects.